CLINICAL TRIAL: NCT00092196
Title: Open-label Extension to: A Randomized, Double-Blind, Parallel-Group Study Conducted Under In-House Blinding Conditions to Determine the Efficacy and Tolerability of Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting Associated With Moderately Emetogenic Chemotherapy
Brief Title: Study of MK0869 for the Prevention of Chemotherapy-Induced Nausea and Vomiting (0869-071)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0869-071 Extension; 2004_064
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Nausea; Vomiting; Breast Neoplasms
Keywords: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting; Breast Neoplasms | interventions — Aprepitant; Duration of Therapy

INTERVENTIONS:
Drug: MK0869, aprepitant / Duration of Treatment: 3 days

SUMMARY:
The purpose of this study is to determine the efficacy and tolerability of an investigational drug for the prevention of chemotherapy-induced nausea and vomiting associated with moderately emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of breast cancer requiring treatment with non-cisplatin moderately emetogenic chemotherapy.
* Patient must have completed participation in the main study for this protocol.

Exclusion Criteria:

* Patient has a central nervous system malignancy.
* Patient will receive radiation to the abdomen or pelvis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2002-12-01 (Actual); Primary Completion 2004-12-01 (Actual); Study Completion 2004-12-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Assessment of adverse experiences using the National Cancer Institute (NCI) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Herrstedt J, Muss HB, Warr DG, Hesketh PJ, Eisenberg PD, Raftopoulos H, Grunberg SM, Gabriel M, Rodgers A, Hustad CM, Horgan KJ, Skobieranda F; Aprepitant Moderately Emetogenic Chemotherapy Study Group. Efficacy and tolerability of aprepitant for the prevention of chemotherapy-induced nausea and emesis over multiple cycles of moderately emetogenic chemotherapy. Cancer. 2005 Oct 1;104(7):1548-55. doi: 10.1002/cncr.21343. PMID 16104039
- [Background] Warr DG, Hesketh PJ, Gralla RJ, Muss HB, Herrstedt J, Eisenberg PD, Raftopoulos H, Grunberg SM, Gabriel M, Rodgers A, Bohidar N, Klinger G, Hustad CM, Horgan KJ, Skobieranda F. Efficacy and tolerability of aprepitant for the prevention of chemotherapy-induced nausea and vomiting in patients with breast cancer after moderately emetogenic chemotherapy. J Clin Oncol. 2005 Apr 20;23(12):2822-30. doi: 10.1200/JCO.2005.09.050. PMID 15837996
- [Derived] Aapro MS, Schmoll HJ, Jahn F, Carides AD, Webb RT. Review of the efficacy of aprepitant for the prevention of chemotherapy-induced nausea and vomiting in a range of tumor types. Cancer Treat Rev. 2013 Feb;39(1):113-7. doi: 10.1016/j.ctrv.2012.09.002. Epub 2012 Oct 11. PMID 23062719
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html